CLINICAL TRIAL: NCT06747793
Title: Evaluation of the Use of Virtual Reality to Reduce Anxiety in Intensive Care Patients
Brief Title: Virtual Reality to Reduce the Anxiety in Critically Ill Patient
Acronym: VRAI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RC31/23/0617
Record Dates: First submitted 2024-11-12; First posted 2024-12-24 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Anxiety; Intensive Care Unit Syndrome
Keywords: Intensive care unit; virtual reality; anxiety; depression; sleep quality
MeSH Terms: conditions — Anxiety Disorders; Depression; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: Clinical interventional trial, randomized, monocentric in the Intensive Care Unit of Toulouse University Hospital.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group: (No Intervention): Standard intensive care unit care without virtual reality stimulation.
- Interventional group: (Experimental): Standard intensive care unit care and 30 minutes of virtual reality stimulation two times per day.
  Interventions: Other: Virtual Reality

INTERVENTIONS:
Other: Virtual Reality — The intervention will consist of relaxing virtual reality stimulation, which will be started after obtaining informed consent. Immersive 360-degree videos (nature environments) will be played inside a head-mounted display, with the video sound played inside headphones. Each virtual reality video will last 30 minutes. The stimulation will be provided two times per day, morning and evening, every day until the patient ICU discharge, or the maximum of 7 days will be reached. The intervention group will also receive standard intensive care unit care, same as in the control group.
  Arms: Interventional group:

SUMMARY:
Anxiety and discomfort generated by repeated medical cares and invasive procedures can induce cognitive disorders in critical illness survivors as post-traumatic stress disorder. For this reason, managing patients' anxiety is particularly important in the intensive care unit. Physicians have recently started using immersive virtual reality (VR), based on real-time interaction with an artificial 360° immersive world, as an adjunctive non-invasive and non-pharmacological anxiolysis technique. The purpose of this project is to assess the virtual reality stimulation to reduce anxiety in Intensive Care Unit (ICU) patients.

DETAILED DESCRIPTION:
Physicians have recently started using immersive VR as an adjunctive non-invasive and non-pharmacological pain control and anxiolysis technique, but the literature on this topic in the adult ICU is quite sparse. In a pilot study, Gerber et al showed the feasibility and acceptance of VR stimulation as a new non-pharmacological intervention to comfort patients during their stay in the ICU and the results appear promising [11]. In our view, the management of anxiety related to healthcare interventions remains a major global challenge and it will be interesting to assess the use of VR in a chronic daily use in the ICU adult patients. Our study will be conducted in the adult intensive care unit of the University of Toulouse, France. All patients who meet the inclusion criteria will be randomized. There will be two distinct groups: the control group will receive standard ICU care, whereas the intervention group will, in addition to the standard ICU care, will receive relaxing VR stimulation two times a day. The intervention will be performed by trained ICU nurses. Anxiety will be assessed by the Visual Analogue Scale for Anxiety (VAS-A) twice by day (morning and evening), sleep quality with the Richards-Campbell Sleep Questionnaire (RCSQ) every morning, depression, and anxiety with the Hamilton Depression Rating Scale (HDRS) and the Hamilton Anxiety Rating Scale (HAM-A) at 3-months after the inclusion. Each patient's heart rate, blood pressure, respiration rate, SatO2, and physical or neurocognitive side effects were used to evaluate if the VR sessions will have any effect on physiology.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient
* Oral consent after free and informed information
* Hospitalized in the multipurpose intensive care unit of Rangueil hospital with an estimated length of stay greater than 24 hours
* Conscious (Glasgow Coma Scale > 8) and Richmond Agitation-Sedation Scale (RASS) sedation score between -1 and +1
* Mechanically ventilated or not
* Person affiliated to or beneficiary of a social security system.

Exclusion Criteria:

* Patient under legal protection (guardianship or curatorship)
* RASS < -1 or > +1
* Visual or hearing difficulties preventing the use of the VR headset
* Severe psychiatric history (severe depression, psychosis, bipolarity), advanced dementia or mental retardation
* Hemodynamic (Norepinephrine support > 0.5 gamma/kg/min) and/or respiratory instability (invasive mechanical ventilation with FiO2 greater than 80%)
* Presence of a malformation or cervical or facial trauma that does not allow the application of the VR headset
* Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Patients' anxiety level after using virtual reality | 7 days
  Visual Analogue Scale for Anxiety (VAS-A) is a scale measuring anxiety from 0 to 100 ; 0: no anxiety, 100: maximum of anxiety

SECONDARY OUTCOMES:
Difference in patient anxiety after using virtual reality | between inclusion and the day 7
  Visual Analogue Scale for Anxiety (VAS-A) variations between inclusion and the day 7. The VAS A is a scale measuring anxiety from 0 to 100 ; 0: no anxiety, 100: maximum of anxiety
Evolution of the psychopathological status: depression | 3 months
  Score to the Hamilton Depression Rating Scale (HDRS) with 16 items from 0 (no symptom) to 4 (high symptom of depression) with a total score from 0 to 30: 0 no depression / 30: depression maximum
Evolution of the psychopathological status: anxiety | 3 months
  Score to the Hamilton Anxiety Rating Scale (HAM-A) with 14 items rom 0 (no symptom) to 4 (high symptom of depression) with a total score from 0 to 56: 0 no anxiety /56: anxiety maximum
Evolution of the Sleep quality | every day through study completion, an average of 5 days
  Score to the Richards-Campbell Sleep Questionnaire (RCSQ) from 0 to 100 (0: worse sleep /100: best sleep
Evaluation of the Safety of using vitural reality in intensive care unit | every day through study completion, an average of 5 days
  Number of side effects that may occur during a VR session
Evaluation of the compliance | 3 months
  Number of virtual reality sessions actually performed by the patient in the intervention group

CONTACTS AND LOCATIONS:
Overall Officials: Floriane PUEL, Dr, Principal Investigator — Hôpital Rangueil, CHU de Toulouse
Locations (1):
- University Hospital of Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No